CLINICAL TRIAL: NCT06305793
Title: RECOVER-AUTONOMIC (IVIG): Randomized Trial of the Effect of IVIG Versus Placebo on Long COVID Symptoms
Brief Title: RECOVER-AUTONOMIC: Platform Protocol, Appendix A (IVIG)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kanecia Obie Zimmerman (Other)
Responsible Party: Sponsor-Investigator, Kanecia Obie Zimmerman, Associate Professor of Pediatrics, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00112597_A; OTA-21-015G (Other: NIH Grant to RTI; RTI subcontracting with DCRI)
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Long COVID; Long Coronavirus Disease 2019 (Covid19); Long Covid-19
Keywords: PASC; POTS
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19 | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Intervention Model Description: In each Appendix trial, each participant will be assigned with equal probability to one of the factorial combinations based on two factors: (1) a study intervention/control and (2) non-pharmacologic intervention/control if the participant is eligible for the study intervention.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- IVIG + Coordinated Care (Experimental): IVIG (Gamunex); 2g /kg monthly for 9 months (36 weeks)
  Interventions: Drug: IVIG (intravenous immunoglobulin); Behavioral: Coordinated Care
- IVIG Placebo + Coordinated Care (Experimental): Saline: Same dosage as IVIG; monthly for 9 months (36 weeks)
  Interventions: Drug: IVIG Placebo; Behavioral: Coordinated Care
- IVIG + Usual Care (Experimental): IVIG (Gamunex); 2g /kg monthly for 9 months (36 weeks)
  Interventions: Drug: IVIG (intravenous immunoglobulin); Behavioral: Usual Care
- IVIG Placebo + Usual Care (Experimental): Saline: Same dosage as IVIG; monthly for 9 months (36 weeks)
  Interventions: Drug: IVIG Placebo; Behavioral: Usual Care

INTERVENTIONS:
Drug: IVIG (intravenous immunoglobulin) — Participants will receive IVIG for 9 months (36 weeks) with a follow-up period for an additional 3 months (total study duration for 12 months).
  Arms: IVIG + Coordinated Care; IVIG + Usual Care
Drug: IVIG Placebo — Normal saline given intravenously will be the control (placebo) product. Blinding IV bag and tubing covers will be used for both IVIG and Placebo.
  Participants will receive placebo for 9 months (36 weeks) with a follow-up period for an additional 3 months (total study duration for 12 months).
  Arms: IVIG Placebo + Coordinated Care; IVIG Placebo + Usual Care
Behavioral: Coordinated Care — Participants will receive coordinated non-pharmacologic care for a duration of 3 months, concurrent with IVIG administration. Coordinated non-pharmacologic care involves volume expansion through high salt diet, water intake, abdominal binder, exercise/rehabilitation, motivation, education, and assisted care through care coordinator.
  Arms: IVIG + Coordinated Care; IVIG Placebo + Coordinated Care
Behavioral: Usual Care — Participants will receive usual non-pharmacologic care (control) for a duration of 3 months, concurrent with IVIG administration.
  Arms: IVIG + Usual Care; IVIG Placebo + Usual Care

SUMMARY:
This study is a platform protocol designed to be flexible so that it is suitable for a wide range of settings within health care systems and in community settings where it can be integrated into COVID-19 programs and subsequent treatment plans.

This protocol is a prospective, multi-center, multi-arm, randomized, controlled platform trial evaluating various interventions for use in the treatment of autonomic dysfunction symptoms, including cardiovascular complications and postural orthostatic tachycardia syndrome (POTS), in Post-Acute Sequelae of SARS-CoV-2 infection (PASC) participants. The interventions tested will include non-pharmacologic care and pharmacologic therapies with study drugs.

DETAILED DESCRIPTION:
The hypothesis is that some of the autonomic dysfunction symptoms are immune-mediated, so immunotherapy and other applicable therapies will result in improvement in autonomic symptoms.

Interventions will be added to the platform protocol as appendices. Each appendix will leverage all elements of the platform protocol, with additional elements described in the individual appendix.

ELIGIBILITY:
Inclusion Criteria:

* See NCT06305780 for RECOVER-AUTO: Platform Protocol level inclusion criteria which applies to this appendix (or sub-study)

Additional Appendix A (IVIG Sub-study) Level Inclusion Criteria:

1. Abnormal active standing test defined as presence of orthostatic tachycardia (an increase of 30 beats per minute (bpm) or more in HR within 10 minutes upon standing without orthostatic hypotension) and experiencing orthostatic symptoms
2. COMPASS-31 Score > 40

Exclusion Criteria:

* See NCT06305780 for RECOVER-AUTO: Platform Protocol level exclusion criteria which applies to this appendix (or sub-study)

Additional Appendix A (IVIG Sub-study) Level Exclusion Criteria:

1. Current or previous IVIG treatment
2. Contraindication to intravenous immunoglobulin.
3. Known allergic reactions to blood products including IVIG and/or subcutaneous immunoglobulin (SCIG), such as history of clinically relevant hemolysis after IVIG infusion, aseptic meningitis, recurrent severe headache, hypersensitivity, severe generalized or severe local skin reactions
4. Selective IgA deficiency
5. Current and recent (within 5 half-lives) use of high-dose corticosteroids (for example for prior solid organ transplant), omalizumab, anti-TNF-alpha inhibitors
6. Use of immunosuppressants such as Plaquenil, or low-dose steroid (prednisone, no more than 10mg a day) will be excluded unless the participant is on stable (>4 weeks) dose
7. Significant thrombotic events after the acute phase of COVID-19 and/or within 6 months of enrollment
8. Veins that are not viable for infusions
9. Not willing to adhere to dosing schedule for IVIG infusions for 9 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2024-03-11 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Orthostatic Hypotension Questionnaire (OHQ)/Orthostatic Intolerance Questionnaire (OIQ) Composite Score | Baseline to End of Intervention (9 months)
  The OHQ / OIQ is a measure of orthostatic intolerance and includes a 6-item symptom assessment (OHSA) and the 4-item Daily Activity Scale (OHDAS). Each item is scored from 0 (none/no interference) to 10 (worst possible/complete interference), describing the preceding week. The OHSA composite score is the average of the first 6 non-zero items and the OHDAS composite score is the average of the last 4 non-zero items. The OHQ/OIQ composite score is the average of the OHSA and OHDAS composite scores. The OHQ/OIQ scales at post-baseline are calculated using only those items that were included in the baseline scores.

SECONDARY OUTCOMES:
Change in Composite Autonomic Symptoms Score 31 (COMPASS-31) | Baseline to End of Intervention (9 months)
  The COMPASS-31 is a patient reported outcome that measures autonomic symptoms across multiple domains commonly seen in patients with PASC. Scores range from 0-100 with higher values representing severe symptoms.
Change in Malmo POTS Symptom Score | Baseline to End of Intervention (9 months)
  The Malmo POTS symptom score assesses symptom burden in postural orthostatic tachycardia syndrome (POTS). It is a self-rating, 12-item score (0-10 per item, total range 0-120) based on patients' own perception of symptoms through visual analogue scale assessment. Higher scores represent more pronounced symptoms.
Change in Active Stand Test | Baseline to End of Intervention (9 months)
  Participants will remain supine for 10 minutes, and data will be acquired at 5 and 10 minutes. Standing test should be performed with HR and BP monitoring at 1, 3, 5 and 10 minutes
Change in blood pressure | Baseline to End of Intervention (9 months)
  measured during Active Stand Test
Change in heart rate (HR) | Baseline to End of Intervention (9 months)
  measured during Active Stand Test
Change in 6-min Walk Test | Baseline to End of Intervention (9 months)
  Normal walking speed will be measured using a standard 6 minute walk
Change in Patient-Reported Outcomes Measurement Information System (PROMIS-29) + 2 Questionnaire | Baseline to End of Intervention (9 months)
  The PROMIS-29 consists of 29 items that assess general domains of health and functioning, including overall physical health, mental health, social health, pain, fatigue, and overall perceived quality of life.
  The PROMIS-29+2 is used to calculate a preference score (PROPr) by the addition of two Cognitive Function Ability items. Scores will be reported as T scores ranging from 0 to 100, with a score of 60 being 1 standard deviation above the mean. Higher scores indicate worse overall health.
Change in step count as measured by a wearable device | Baseline to End of Intervention (9 months)
  measured by activity tracker
Change in heart rate as measured by a wearable device | Baseline to End of Intervention (9 months)
  measured by activity tracker
Proportion of participants who experience individual (SAEs | Baseline to Follow-up (12 months)
  These will be analyzed in the safety population.
Proportion who experience any one or more ( Serious Adverse Event) SAEs | Baseline to Follow-up (12 months)
  These will be analyzed in the safety population.
Incidence of SAEs leading to discontinuation | Baseline to Follow-up (12 months)
  These will be analyzed in the safety population.
Incidence of Events of Special Interest (ESIs) | Baseline to Follow-up (12 months)
  Each study drug may have a unique list of ESIs

OTHER OUTCOMES:
Changes in Autonomic Function Testing | Baseline to End of Intervention (9 months)
  * Head-up tilt (HUT) test
  * Valsalva maneuver with a pressure of 40 mmHg for 15 seconds
  * Deep breathing test
  * Skin biopsy (if applicable as per Appendix)
  * Transcranial doppler (TCD), if available
Change in Vanderbilt Orthostatic Symptoms Score (VOSS) | Baseline to End of Intervention (9 months)
  The VOSS consists of 9 orthostatic symptoms rated on a scale of 0 (no symptom) to 10 (worst the participant has experienced) at the end of each Head-up Tilt test. Scores range from 0-90 with higher scores representing worse symptoms.
Change in PASC Symptom Questionnaire | Baseline to End of Intervention (9 months)
  Participants will be asked to complete a questionnaire that asks about the presence of PASC symptoms. This questionnaire includes additional PASC symptoms that are not directly related to autonomic dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Grainger, MD, Study Chair — Duke Clinical Research Institute; Cyndya Shibao, MD, Study Chair — Vanderbilt University Medical Center; Peter Novak, MD, Study Chair — Harvard; Pam Taub, MD, Study Chair — University of California, San Diego; Tae Chung, MD, Study Chair — Johns Hopkins University
Locations (1):
- All sites listed under NCT06305780, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
The summary of results will be shared on the study website: https://recovercovid.org/

REFERENCES:
- See also: Related Info — http://recovercovid.org/

DOCUMENTS (1):
  • Informed Consent Form (2024-01-15): https://cdn.clinicaltrials.gov/large-docs/93/NCT06305793/ICF_000.pdf